CLINICAL TRIAL: NCT01039480
Title: Aspirin- and Clopidogrel-Resistance: Non-compliance and Other Contributing Factors
Brief Title: Aspirin and Clopidogrel Resistance Study
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Philipp N. Walter, Investigator, Pharmaceutical Care Research Group
Other Study IDs: PCRG_003_PW
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Drug Resistance
Keywords: pharmacological biomarker; compliance monitoring; platelet aggregometry; resistance; Platelet Aggregation Inhibitors; Medication Non-Compliance
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood samples for routine laboratory testing and platelet aggregometry blood samples for pharmacogenetic analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- dual therapy (ASS/CLO): patients with a prescription for dual antiplatelet therapy with aspirin AND clopidogrel
- clopidogrel users (CLO): patients with a prescription for clopidogrel
- aspirin users (ASP): patients with a prescription for aspirin

SUMMARY:
Resistance to antiplatelet drugs (aspirin, clopidogrel) is a recognized phenomenon with a prevalence from 17% to 35%. Resistance as detected by in vitro tests such as Multiple Electrode Aggregometry (MEA) has been shown to predict clinical therapy failure. Resistance can be caused by clinical, cellular and pharmacogenetic factors. Non compliance is suspected to be an important contributing factor. In this study, compliance will be assured with an electronical compliance monitoring system. Factors to non response will be identified to find plausible explanations when in vitro platelet aggregation inhibition is insufficient despite assured compliance. This study will help to disclose the relationship between compliance, biomarker and clinical outcome as well as to quantify the impact of non compliance to the resistance phenomenon as measured by MEA.

ELIGIBILITY:
Inclusion Criteria:

* Patients prescribed aspirin and/or clopidogrel for both including both cardiovascular and cerebrovascular indications seeing their general practitioner in or nearby Olten/SO for any medical purpose
* Patients with oral and written German language ability

Exclusion Criteria:

* Patients living in care homes
* Patients not preparing their drugs on their own (e.g. outpatient medical assistance through "spitex").
* Patients with acute cardiac symptoms

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a prescription for aspirin and/or clopidogrel seeing their general practitioner (GP) for any purpose
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2010-05; Primary Completion 2011-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Platelet aggregation, initial and after one week under compliance monitoring. | 1 week

SECONDARY OUTCOMES:
Data on compliance (measured by electronic compliance monitoring, Morisky MMAS-8 and BMQ Score) | 1 week
Frequency of contributing factors to non-response in responders compared to non-responders (pharmacogenetics, clinical factors and drug-drug interactions) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kurt E Hersberger, PhD, Study Chair — Pharmaceutical Care Research Group, Departement of Pharmacy, University Basel; Michel Romanens, MD, Principal Investigator — Kardiologische Praxis, Olten/SO; Dimitrios Tsakiris, MD, Study Director — Hemostaseology Lab, University Hospital Basel; Philipp N Walter, MSc, Principal Investigator — Pharmaceutical Care Research Group, Department of Pharmacy, University of Basel
Locations (1):
- Study Centre at Aarelab AG, Olten, Olten, Canton of Solothurn, Switzerland

REFERENCES:
- [Derived] Walter PN, Tsakiris DA, Romanens M, Arnet I, Hersberger KE. Antiplatelet resistance in outpatients with monitored adherence. Platelets. 2014;25(7):532-8. doi: 10.3109/09537104.2013.845743. Epub 2013 Oct 31. PMID 24175592
- See also: Pharmaceutical Care Research Group, Departement of Pharmacy, University Basel — http://www.pharmacare.unibas.ch